CLINICAL TRIAL: NCT01194479
Title: The Effect of the Beta 2 Agonist, Formoterol, on Recovery From Hypoglycemia
Brief Title: Effect of Formoterol on the Counterregulatory Hormonal Response to Hypoglycemia in Type 1 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HIC1005006832; R37-20495 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; hypoglycemia; formoterol
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 1 Diabetics (Active Comparator): The active group were participants with type 1 diabetes.
  Interventions: Drug: Formoterol; Other: Placebo
- Healthy Volunteers (Other): The control group were participants without diabetes, matched by sex, age and BMI to the active comparator group.
  Interventions: Drug: Formoterol; Other: Placebo

INTERVENTIONS:
Drug: Formoterol — Formoterol inhaler, 12mcg capsules, 4 capsules for one administration
  Other Names: Foradil Aerolizer
Other: Placebo — Participants in both arms received placebo on 1 of the 2 visits.

SUMMARY:
Insulin treatment often causes the blood glucose levels to fall too low. The body usually responds to low blood glucose levels by releasing hormones which act against the insulin to help correct the low blood glucose levels. However, this hormone response can be altered in people with diabetes. Currently there are no therapeutic agents that can be used to improve the recovery from hypoglycemia (low blood sugar). The aim of this study is to determine whether a formoterol inhaler can be used to improve and accelerate the recovery from hypoglycemia in patients with type 1 diabetes.

DETAILED DESCRIPTION:
Note: Below is the original detailed description submitted in 2010. The recruitment for this study was stopped at 7 subjects in each study arm. The study design and outcome measures did not change for this study. See below for further details.

Original: 15 subjects with well controlled type 1 diabetes and regular hypoglycemia and 15 healthy volunteers will be recruited for this study.

If you agree to participate in this study, you will be asked to participate in a screening at Yale New Haven Hospital. Each study subject will undergo two hypoglycemic clamp studies (a procedure where the blood sugar is closely regulated with intravenous insulin and glucose.) In these hypoglycemic clamp studies, the subject will be given an inhaler. On one visit the inhaler will contain formoterol capsules and on the other visit, the subject will be given 'dummy' capsules. Subjects will be required to be admitted to the HRU the night before the study so that glucose levels can be stabilized and hypoglycemia avoided.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes (well controlled, 2-3 hypoglycemic episodes/wk)
* age 18-50
* BMI 18-30

Exclusion Criteria:

* pregnancy
* significant diabetes complications
* liver disease, cirrhosis
* cardiac disease
* neurological disorder
* autonomic neuropathy
* kidney disease
* lactose intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Result] Belfort-DeAguiar RD, Naik S, Hwang J, Szepietowska B, Sherwin RS. Inhaled Formoterol Diminishes Insulin-Induced Hypoglycemia in Type 1 Diabetes. Diabetes Care. 2015 Sep;38(9):1736-41. doi: 10.2337/dc14-2472. Epub 2015 Jul 7. PMID 26153273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects and Type 1 Diabetics were recruited to participate in the study. Subjects in either arm were randomized to receive a placebo or the study drug: Formoterol in either the first or second visit.
Groups:
- Control: Placebo: Healthy volunteers that received Placebo first, the Formoterol.
- Control: Formoterol: Healthy volunteers that received Formoterol first, then Placebo.
- Type 1 Diabetics: Placebo: Type 1 Diabetics that received Placebo first, then Formoterol.
- Type 1 Diabetics: Formoterol: Type 1 Diabetics that received Formoterol first, then Placebo.
Period: Overall Study
Arm/Group | Control: Placebo | Control: Formoterol | Type 1 Diabetics: Placebo | Type 1 Diabetics: Formoterol
Started | 3 | 4 | 2 | 5
Cross-over at Second Visit | 3 | 4 | 2 | 5
Completed | 3 | 4 | 2 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Type 1 Diabetics | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8) | 31 (11) | 33.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 3 | 6
Body Mass Index (BMI, kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (2.1) | 25.8 (2.9) | 24.8 (2.7)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 70.0 (12.9) | 70.2 (10.6) | 70.1 (11.3)
HbA1c (%) [Mean (Standard Deviation); unit: %] | 5.3 (2.6) | 6.8 (2.6) | 6.1 (1.0)
HbA1c (mmol/mol) [Mean (Standard Deviation); unit: mmol/mol] | 34.5 (2.6) | 51.3 (8.5) | 43.5 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Glucagon (pg/mL)
Description: Glucagon levels will be measured throughout the study to assess whether there are changes during hypoglycemia with inhaled formoterol. These levels will be checked every 20 minutes during the 120 minute study session. Results are presented at the Basal, Euglycemia (30 minutes) and Hypoglycemia (105-120 minutes) stages.
Time Frame: up to 120 minutes
Population: Results are pooled at the arm level and split by placebo and control regardless of randomization order.
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Control: Placebo: Healthy volunteers that received Placebo on the first or second visit.
- Control: Formoterol: Healthy volunteers that received Formoterol on the first or second visit.
- Type 1 Diabetics: Placebo: Type 1 Diabetics that received placebo on the first or second visit.
- Type 1 Diabetics: Formoterol: Type 1 Diabetics that received Formoterol on the first or second visit.
Arm/Group | Control: Placebo | Control: Formoterol | Type 1 Diabetics: Placebo | Type 1 Diabetics: Formoterol
Number analyzed (Participants) | 7 | 7 | 7 | 7
pg/mL
  Basal | 76 (13) | 74 (11) | 53 (8) | 56 (10)
  Euglycemia | 59 (11) | 58 (13) | 55 (10) | 54 (9)
  Hypoglycemia | 66 (16) | 73 (18) | 43 (8) | 46 (9)

2. Secondary Outcome: Blood Glucose Levels (Average)
Description: Blood glucose levels will be checked every 5 minutes during the 120 minute study session in order to maintain blood glucose levels in the normal and hypoglycemic range. Presented is the average of the collected values.
Time Frame: Up to 120 minutes
Population: Subjects are pooled across randomized conditions in their respective study arms and reported overall.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control: Placebo | Control: Formoterol | Type 1 Diabetics: Placebo | Type 1 Diabetics: Formoterol
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 57.38 (3.45) | 58.39 (2.40) | 53.21 (2.57) | 55.43 (4.40)

3. Primary Outcome: Epinephrine (pg/mL)
Description: Epinephrine levels will be measured throughout the study to assess whether there are changes during hypoglycemia with inhaled formoterol. These levels will be checked every 20 minutes during the 120 minute study session. Results are presented at the Basal, Euglycemia (30 minutes) and Hypoglycemia (105-120 minutes) stages
Time Frame: up to 120 minutes
Population: Results are pooled at the arm level and split by placebo and control regardless of randomization order.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Control: Placebo | Control: Formoterol | Type 1 Diabetics: Placebo | Type 1 Diabetics: Formoterol
Number analyzed (Participants) | 7 | 7 | 7 | 7
pg/mL
  Basal | 15 (4) | 16 (5) | 18 (4) | 17 (5)
  Euglycemia | 12 (3) | 12 (4) | 21 (5) | 13 (2)
  Hypoglycemia | 46 (15) | 55 (22) | 44 (15) | 19 (4)

4. Primary Outcome: Norepinephrine (pg/mL)
Description: Norepinephrine levels will be measured throughout the study to assess whether there are changes during hypoglycemia with inhaled formoterol. These levels will be checked every 20 minutes during the 120 minute study session. Results are presented at the Basal, Euglycemia (30 minutes) and Hypoglycemia (105-120 minutes) stages
Time Frame: up to 120 minutes
Population: Results are pooled at the arm level and split by placebo and control regardless of randomization order.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Control: Placebo | Control: Formoterol | Type 1 Diabetics: Placebo | Type 1 Diabetics: Formoterol
Number analyzed (Participants) | 7 | 7 | 7 | 7
pg/mL
  Basal | 185 (37) | 192 (24) | 180 (28) | 133 (13)
  Euglycemia | 216 (31) | 273 (22) | 226 (31) | 211 (30)
  Hypoglycemia | 156 (21) | 181 (14) | 241 (30) | 190 (32)

ADVERSE EVENTS:
Time Frame: Adverse events are reported by the study arm and randomized visit order.
Groups:
- Control: Placebo: Healthy volunteers that received Placebo on the first visit.
- Control: Formoterol: Healthy volunteers that received Formoterol on the first visit.
- Type 1 Diabetics: Placebo: Type 1 Diabetics that received placebo on the first visit.
- Type 1 Diabetics: Formoterol: Type 1 Diabetics that received Formoterol on the first visit.
Arm/Group | Control: Placebo | Control: Formoterol | Type 1 Diabetics: Placebo | Type 1 Diabetics: Formoterol
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 3/7 | 0/7 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control: Placebo (N=7) | Control: Formoterol (N=7) | Type 1 Diabetics: Placebo (N=7) | Type 1 Diabetics: Formoterol (N=7)
Shakiness (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hunger (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tiredness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mild Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Light Headedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes